CLINICAL TRIAL: NCT05474014
Title: Investigation of the Effectiveness of Superior Trunk Block Applied for Upper Arm Surgery Operation Analgesia
Brief Title: Superior Trunk Block Applied for Upper Arm Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Korgün Ökmen, Assoc.Phd.M.D, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/06-12
Record Dates: First submitted 2022-07-19; First posted 2022-07-26 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- superior trunk block (Active Comparator): Ultrasound guided superior trunk block with 10 ml % 0.25 bupivacaine
  + 400 mg tramadol, IV 4 mg/ mL tramadol solution into 100 mL normal saline; PCA (patient-controlled analgesia): 0.3 mg/kg bolus, 10 mg Demand dose and 20 min lock out interval, six-hour limit infusion to attain 100 mg. Maximum daily dose was set at 400 mg.
  Interventions: Procedure: superior trunk block; Drug: intravenous patient-controlled analgesia
- tramadol (Active Comparator): 400 mg tramadol, IV 4 mg/ mL tramadol solution into 100 mL normal saline; PCA (patient-controlled analgesia): 0.3 mg/kg bolus, 10 mg Demand dose and 20 min lock out interval, six-hour limit infusion to attain 100 mg. Maximum daily dose was set at 400 mg.
  Interventions: Drug: intravenous patient-controlled analgesia

INTERVENTIONS:
Procedure: superior trunk block — Local anesthetic injection will be applied to the superior trunk of the brachial plexus accompanied by ultrasonography.
  Arms: superior trunk block
Drug: intravenous patient-controlled analgesia — Analgesics will be given using a patient-controlled analgesia device.

SUMMARY:
Nerve blocks applied with ultrasonography are currently used for many post-operative pain and operations. Providing adequate area analgesia is the primary goal of clinicians, as early mobilization is suggested after shoulder and arm surgery.

In this study aimed to investigate the effect of superior trunk block application on postoperative analgesic and motor functions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were in the American Society of Anesthesiologists (ASA) I-III class
* Underwent upper arm surgery

Exclusion Criteria:

* Previous local anesthetic allergy,
* Having a bleeding diathesis disorder,
* Mental disorder,
* Allergic to the drugs used,
* Patients who did not consent to participate in the study,
* Presence of infection in the block area,
* Patients with a body mass index above 30

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Postoperative 24 hours
  Visual Analog Scale was used for pain.Pain intensity was measured using 0-10 cm visual analogue scale (VAS). (0=no pain, 10=intolerable pain)

SECONDARY OUTCOMES:
tramadol consumption amount | Postoperative 24 hours
  tramadol consumption amount with patient-controlled analgesia device
additional analgesic use amount | Postoperative 24 hours
  The amount of paracetamol (intravenous, 1 g) or non-steroidal anti-inflammatory drug to be administered to patients with a Visuel analog scale above 5 after the operation.
postoperative complications | Postoperative 24 hours
  shortness of breath, hiccups, hoarseness
Horner syndrome | Postoperative 24 hours
  Horner syndrome is a rare condition classically presenting with partial ptosis (drooping or falling of upper eyelid), miosis (constricted pupil), and facial anhidrosis (loss of sweating) due to a disruption in the sympathetic nerve supply

CONTACTS AND LOCATIONS:
Overall Officials: Korgün Ökmen, Assoc. PhD., Principal Investigator — Sağlık Bilimleri Üniversitesi Bursa Yüksek İhtisas Eğitim Ve Araştırma Hastanesi
Locations (1):
- Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Turkey (Türkiye)